CLINICAL TRIAL: NCT03071523
Title: Clinical and Radiographic Comparison of Coronally Advanced Lingual Flap to Periosteal Releasing Incision for Flap Advancement in Partially Edentulous Patients Undergoing Guided Bone Regeneration Using Titanium Mesh: RCT.
Brief Title: Flap Advancement Techniques in Ridge Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rasha Attia, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-2017-01-130
Record Dates: First submitted 2017-01-13; First posted 2017-03-07 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Flap Advancement; Primary Wound Closure

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- coronally advanced lingual flap (Experimental): Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side. On the buccal side, full thickness mucoperiosteal flap will be raised with horizontal incision 1-3 mm in depth performed in the buccal flap. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. A band of mylohyoid muscle is inserted into the inner part of the lingual flap approximately 5 mm from the crest in an apical direction. A blunt instrument will be inserted below that connective band, and, with gentle traction in the coronal direction, this muscular insertion should be detached freeing the lingual flap from the mylohyoid.
  Interventions: Procedure: coronally advanced lingual flap
- periosteal releasing incision technique (Active Comparator): Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side and a full thickness flap will be raised. Xenograft and Ti-mesh will be used to augment the defective site then incremental incisions of 1-3 mm into the periosteum and submucosa will be used to advance the muco-periosteal flap. The flap will then be sutured with interrupted sutures.
  Interventions: Procedure: periosteal releasing incision

INTERVENTIONS:
Procedure: coronally advanced lingual flap — Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side. On the buccal side, full thickness mucoperiosteal flap will be raised with horizontal incision 1-3 mm in depth performed in the buccal flap. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. A band of mylohyoid muscle is inserted into the inner part of the lingual flap approximately 5 mm from the crest in an apical direction. A blunt instrument will be inserted below that connective band, and, with gentle traction in the coronal direction, this muscular insertion should be detached freeing the lingual flap from the mylohyoid.
  Arms: coronally advanced lingual flap
Procedure: periosteal releasing incision — Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side and a full thickness flap will be raised. Xenograft and Ti-mesh will be used to augment the defective site then incremental incisions of 1-3 mm into the periosteum and submucosa will be used to advance the muco-periosteal flap. The flap will then be sutured with interrupted sutures.
  Arms: periosteal releasing incision technique

SUMMARY:
Different augmentation techniques has been proposed to resolve problem of hard and/or soft tissue ridge defects to enable dental implant placement. Guided bone regeneration GBR procedure is considered as an acceptable reliable surgical procedure for localized ridge augmentation. Exposure of the membrane used for the GBR is considered a major disadvantage of this procedure. In order to avoid such complication, various flap advancement techniques have been proposed such as Periosteal releasing incision,Double-Flap Incision,Coronally advanced lingual flap. The study compare between the flap advancement provided by Periosteal releasing incision,versus,Coronally advanced lingual flap in the treatment of class 1 ridge defect.

DETAILED DESCRIPTION:
Two arms RCT will be conducted as followed:

Group A (intervention):

Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side. On the buccal side, full thickness mucoperiosteal flap will be raised with horizontal incision 1-3 mm in depth performed in the buccal flap. On the lingual side, a full-thickness mucoperiosteal flap will be elevated until reaching the mylohyoid line. A band of connective tissue continuing with the epimysium of the mylohyoid muscle is usually located in the first molar area, and is1 to 2 cm wide in a mesiodistal direction. This band is inserted into the inner part of the lingual flap approximately5 mm from the crest in an apical direction. A blunt instrument will be inserted below that connective band, and, with gentle traction in the coronal direction, this muscular insertion should be detached freeing the lingual flap from the mylohyoid muscle. Then Xenograft and Ti-mesh will be used to augment the defective site and the flap will then be sutured with interrupted sutures.

Group B ( control ):

Full-thickness crestal incision will be made over the edentulous ridge followed by one full-thickness vertical incision on the buccal side and a full thickness flap will be raised. Xenograft and Ti-mesh will be used to augment the defective site then incremental incisions of 1-3 mm into the periosteum and submucosa will be used to advance the muco-periosteal flap. The flap will then be sutured with interrupted sutures.

ELIGIBILITY:
Inclusion Criteria:

* Partially edentulous patients in the mandibular posterior region.
* Patients with healthy systemic conditions.
* Insufficient ridge width (< 5mm).
* Presence of proper inter-arch space for placement of the implant prosthetic part with adequate soft tissue biotype (≥ 2mm).
* No clinical evidence of active periodontal disease or oral infections.

Exclusion Criteria:

* Patients with systemic conditions that may interfere with the results of the study.
* Patients with local pathological defects related to the area of interest.
* Unmotivated, uncooperative patients with poor oral hygiene.
* Patients with habits that may jeopardize the implant longevity and affect the results of the study such as smoking, alcoholism or para-functional habits.
* History of bone associated diseases or medication affecting bone metabolism e.g. bisphosphonate treatment.
* History of radiation therapy in the head or neck region.
* Current antitumor chemotherapy.
* Pregnancy.
* Inflammatory and autoimmune diseases of the oral cavity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-12-20 (Actual)

PRIMARY OUTCOMES:
Flap advancement | Intra-operative after flap release by either periosteal releasing incision or lingual flap advancment
  Using periodontal probe in millimeters.

SECONDARY OUTCOMES:
Bone width gain | 9 month
  Using Cone Bean Computed tomography in millimeters.
Postoperative membrane exposure | 9 month
  Using periodontal probe in millimeters.
Postoperative Pain | 2 weeks
  VAS scale
Postoperative swelling | 2 weeks
  VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Manal M. Hosny, Professor, Study Chair — Cairo University; Hany E. El-Nahas, Assist. Prof, Study Director — Cairo University
Locations (1):
- Rasha Attia, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No